CLINICAL TRIAL: NCT07197814
Title: Evaluation of the Hypoallergenicity of a New Formula Based on Hydrolyzed Rice Proteins in Children With IgE-mediated Cow's Milk Allergy
Brief Title: Evaluation of the Tolerance of a New Formula Based on Hydrolyzed Rice Proteins in Children With Cow's Milk Allergy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health and Happiness Research Limited (Industry)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: BST-001
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: IgE-Mediated Cow Milk Allergy
Keywords: Cow's milk allergy; Hydrolyzed rice proteins-based formula; IgE-mediated; Oral food challenge; Hypoallergenicity; Tolerance
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBPCFC = Day 1: Rice formula; Day 2: Placebo formula (Experimental): On Day 1 of the DBPCFC, subjects will receive the Rice formula. On Day 2 of the DBPCFC, subjects will receive the Placebo formula. If subjects tolerate the Rice formula during this DBPCFC, they will then be fed the Rice formula for 7 days.
  Interventions: Other: Rice formula (New formula based on hydrolysed rice proteins); Other: Placebo formula
- DBPCFC = Day 1: Placebo formula; Day 2: Rice formula (Experimental): On Day 1 of the DBPCFC, subjects will receive the Placebo formula. On Day 2 of the DBPCFC, subjects will receive the Rice formula. If subjects tolerate the Rice formula during this DBPCFC, they will then be fed the Rice formula for 7 days.
  Interventions: Other: Rice formula (New formula based on hydrolysed rice proteins); Other: Placebo formula

INTERVENTIONS:
Other: Rice formula (New formula based on hydrolysed rice proteins) — Infant formula based on hydrolysed rice proteins.
Other: Placebo formula — The placebo formula will be the formula the subject is currently successfully fed with as part of his/her diet to eliminate cow's milk proteins.

SUMMARY:
The goal of this clinical trial is to see if a new formula based on hydrolysed rice proteins (Rice formula) is well tolerated by infants and young children with cow's milk allergy. In case the Rice formula is well tolerated, the formula will be considered " hypoallergenic ".

The main question it aims to answer is: Does the Rice formula cause allergic reactions in infants and young children who are allergic to cow's milk? Researchers will compare during a double-blind placebo-controlled food challenge (DBPCFC) the Rice formula to a Placebo formula to see if any allergic symptom appears after feeding with the Rice formula. If children do not show any allergic symptoms during the DBPCFC, they will then be exclusively formula-fed the Rice formula for 7 days.

Participants will:

* come at the hospital twice (around 7 days apart) for the DBPCFC
* then, after this procedure, be fed the Rice formula for 7 days, as a replacement for their usual infant formula

Their parents will pay attention to the appearance of any allergic symptom after each day of the DBPCFC, and during the 7-day feeding period. They will keep a diary of any adverse event in their child, the use of any concomitant treatment, and the introduction in their child's diet of any new allergenic food. In addition, during the 7-day feeding period, they will report quantities of the Rice formula consumed, data on regurgitations/vomiting if any, stool consistency/frequency/colour and their satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Infants and young children between 1 and 36 months of age
* Consuming at least 240 ml/day of formula
* Gestational age ≥ 37 weeks
* Diagnosis of IgE-mediated CMA confirmed through a DBPCFC performed within 3 months prior to the enrolment
* Stable clinical condition and free from any symptoms possibly related to CMA for at least ≥4 weeks prior to recruitment
* Observing a strict cow's milk proteins elimination diet for at least 4 weeks prior to study enrollment
* Parents or legal guardians agree not to enroll infant in another interventional clinical study while participating in this study
* Written informed consent form obtained from both parents (or legally acceptable representative [LAR], if applicable)
* Infant's parents / LAR are of legal age of majority, must have parental authority, must understand the informed consent form and other study documents, and are willing and able to fulfill the requirements of the study protocol.
* Signed authorization obtained from both parents or legal guardian to use and/or disclose Protected Health Information for infant from birth through the length of the study period

Exclusion Criteria:

* Infant is exclusively breastfed.
* Any chronic diseases, chromosomal or major congenital anomalies (based on medical history and/or commonly performed diagnostic criteria).
* Major gastrointestinal disease/abnormalities (other than CMA).
* Other food allergies
* Eosinophilic disorders of the gastrointestinal tract.
* Evidence of non-IgE-mediated CMA.
* Immunodeficiency.
* Use of drugs that may interfere with the interpretation and safety of the SPT procedure planned on Inclusion visit such as antihistamines and topical corticosteroids in the previous week, angiotensin-converting enzyme (ACE) inhibitors within the 2 days before or beta-blockers the day before as well as skin moisturizers used on the skin where solution drops will be applied.
* Previous use of systemic immunomodulatory treatment at any time before study entry.
* Use of systemic antibiotics or anti-mycotic drugs within 4 weeks before study entry.
* Persistent wheeze or chronic respiratory disease.
* Severe uncontrolled eczema.
* Currently participating or having participated in another interventional clinical study within 4 weeks prior to enrollment.
* Infant's parents/LAR have medical or psychiatric condition that, in the judgement of the Investigator, would make the subject inappropriate for entry into the study.

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Hypoallergenicity of the Rice formula | At the end of the 7-day open feeding period
  It will be assessed through the absence of medically confirmed allergic reaction to the study formula (Rice formula), based on assessment of clinical signs and symptoms at clinical DBPCFC testing and during the 7-day open feeding period.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II, University of Naples, Department of Translational Medical Science, Napoli, Italy